CLINICAL TRIAL: NCT04018300
Title: Assessment of Gastrointestinal Symptoms and Other Side Effects After Three Week Oral Ferrous Sulfate and Iron-enriched Aspergillus Oryzae Supplementation in Young Female Subjects
Brief Title: Iron Supplementation and Side Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Dr. Manju B. Reddy, Professor, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SEAS
Record Dates: First submitted 2019-05-03; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Iron Deficiency Anemia; Iron Overload
Keywords: ferrous sulfate; non-transferrin bound iron; oral iron supplement; oral iron supplement side effects
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Overload | interventions — ferrous sulfate; Starch

STUDY DESIGN:
Intervention Model Description: Three armed, cross-over, double blinded design. Fifteen subjects will be randomized to treatment FeSO4, ASP or placebo for two week per treatment. Following each treatment, will be a two week washout period whereby subjects will not consume a supplement. Baseline and final blood draws of each treatment will be collected, in addition to serum collection at 0h, 1h, 2h, 3h, 4h following one dose to determine NTBI concentration curve.
Who Masked: Participant, Investigator
Masking Description: Treatments will be randomized to A or B. Investigators will be blinded to the corresponding treatment, in addition to the subjects being randomized to follow the sequence of supplements as ACB or BCA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ferrous sulfate (Experimental): Subjects will take a 65 mg Fe capsule of ferrous sulfate, once daily for 21 consecutive days. The first treatment capsule will be consumed with a semi-purified meal (egg albumin, sugar, vanilla, maltodextrose and corn oil) and will have blood drawn hours 0, 1, 2, 3, 4, 6 and 8 post consumption. Serum will be used to determine non-transerrin bound iron, serum iron and percent saturation. Throughout the treatment period, subjects are informed to consume the capsule with food and report symptoms in an online questionnaire. Following three weeks treatment, participants return for a blood draw and oxidative stress indicators are measured. A three week washout period with placebo treatment takes place between treatment crossover.
  Interventions: Dietary Supplement: Ferrous sulfate
- Aspiron (Experimental): AspironTM which is an iron-enriched supplement will follow the same guidelines and protocol as ferrous sulfate arm. Equivalent 65 mg Fe per capsule will be administered to participants.
  Interventions: Dietary Supplement: Aspiron
- Placebo (Placebo Comparator): Participants will follow the same description for the other two experimental treatment groups. Capsules will be given to subjects in opaque formation, therefore will be unable to differentiate the iron supplements.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ferrous sulfate — 65 mg Fe as ferrous sulfate
  Arms: Ferrous sulfate
Dietary Supplement: Aspiron — 65 mg Fe as iron-enriched koji culture, called AspironTM
  Other Names: Aspergillus oryzae
  Arms: Aspiron
Other: Placebo — Contains maltodextrin.
  Other Names: Starch pill
  Arms: Placebo

SUMMARY:
The objective of this study is to examine patient-reported gastrointestinal side effects, as well as iron status indicators, inflammatory markers and oxidative stress following administration of ferrous sulfate and iron-enriched Aspergillus oryzae supplementation.

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) afflicts more than 2 billion people globally, making it the most prevalent nutrient disorder, today. Inadequate dietary intake of iron results in consequences like cognitive decline, fatigue, abnormal growth and adverse pregnancy outcomes. These ramifications have associated burdens on economical progression due to decreased market productivity. Inorganic iron supplements like ferrous sulfate (FeSO4) are most commonly used to treat IDA, however known associated side effects occur, decreasing compliancy in individuals. Moreover, inorganic iron salts present a large bolus of iron to the intestinal lumen, resulting in non-transferrin bound iron which leads to systemic inflammation and further exacerbation of chronic diseases. Organic iron compounds have strong potential to be utilized for supplementation, however only under circumstances in which contain high absorbance. Seventeen subjects were randomized in a three-armed, double-blinded crossover design to examine the differences among three treatments (FeSO4, ASP-s and placebo). Outcomes will be to assess acute inflammatory proteins, oxidative stress, iron status indicators, non-transferrin bound iron and gastrointestinal-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* Female
* BMI < 30 kg/m2
* Nonsmoker
* Non pregnant
* Non lactating
* No food allergies to wheat or dairy
* No history of gastrointestinal diseases/disorders
* Willing to discontinue use of vitamin/mineral supplements
* No medications that interfere with iron absorption
* No blood or plasma donations during study period

Exclusion Criteria:

* History of gastrointestinal diseases or disorders
* Donating blood or plasma two weeks prior to study period
* On medications interfering with iron absorption
* Food allergies to wheat or dairy
* Pregnant or lactating
* Smoker
* Anemic (< 120 g/L)
* Ferritin > 40 ug/L

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Area under the serum iron curve over 8 hours | 0,1,2,3,4,6 and 8 hours
  Serum iron concentrations (µM) measured over 8 hours following consumption of either Ultimine, FeSO4, or placebo capsules at baseline (0h).
Area under the NTBI curve over 8 hours | 0,1,2,3,4,6 and 8 hours
  NTBI (µM) concentrations measured over 8 hours following consumption of either Ultimine, FeSO4, or placebo capsules at baseline (0h).
Area under the percent transferrin saturation curve over 8 hours | 0,1,2,3,4,6 and 8 hours
  Percent transferrin (%) saturation concentrations measured over 8 hours following consumption of either Ultimine, FeSO4, or placebo capsules at baseline (0h).

SECONDARY OUTCOMES:
Change in protein carbonyls | Baseline and 21 days
  Change from baseline to 21 days of protein carbonyls (nmol/mL) oxidative stress after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in thiobarbituric acid reactive substances (TBARS) | Baseline and 21 days
  Change from baseline to 21 days of TBARS (µM) oxidative stress after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in hepcidin | Baseline and 21 days
  Change from baseline to 21 days of inflammatory status via hepcidin (ng/mL) after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in C-reactive protein | Baseline and 21 days
  Change from baseline to 21 days of inflammatory status via C-reactive protein (mg/L) after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in serum ferritin | Baseline and 21 days
  Change from baseline to 21 days of iron status through serum ferritin (µg/L) after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in hemoglobin | Baseline and 21 days
  Change from baseline to 21 days of iron status through hemoglobin (g/dL) production after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in hematocrit | Baseline and 21 days
  Change from baseline to 21 days of iron status through hematocrit (%) production after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in soluble transferrin receptor (sTFR) | Baseline and 21 days
  Change from baseline to 21 days of iron status through sTFR (ng/mL) production after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in total iron binding capacity (TIBC) | Baseline and 21 days
  Change from baseline to 21 days of iron status through TIBC (µg/dL) production after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in glomerular filtration rate (eGFR) | Baseline and 21 days
  Change from baseline to 21 days of kidney function through eGFR (mL/min/1.73m2) production after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in creatinine | Baseline and 21 days
  Change from baseline to 21 days of kidney function through creatinine (mg/dL) production after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in blood urea nitrogen (BUN) | Baseline and 21 days
  Change from baseline to 21 days of kidney function through BUN (mg/dL) production after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in aspartate aminotransferase (AST) | Baseline and 21 days
  Change from baseline to 21 days of kidney function through AST (U/L) production after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Change in alanine aminotransferase (ALT) | Baseline and 21 days
  Change from baseline to 21 days of kidney function through ALT (U/L) production after taking either Ultimine, FeSO4, or placebo for 3 consecutive weeks.
Gastrointestinal symptoms | 21 days
  Symptoms questionnaire was distributed 3 days/week over 3 weeks/treatment. Total survey per supplemental treatment included 9 surveys. Participants described how the supplement contributed to gastrointestinal distress, such as, constipation, diarrhea, fatigue, abdominal discomfort, nausea, headaches, and heartburn.

CONTACTS AND LOCATIONS:
Overall Officials: Manju B Reddy, PhD, Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Publication in a journal

REFERENCES:
- [Derived] Bries AE, Wang C, Agbemafle I, Wels B, Reddy MB. Assessment of Acute Serum Iron, Non-Transferrin-Bound Iron, and Gastrointestinal Symptoms with 3-Week Consumption of Iron-Enriched Aspergillus oryzae Compared with Ferrous Sulfate. Curr Dev Nutr. 2019 Nov 7;3(12):nzz127. doi: 10.1093/cdn/nzz127. eCollection 2019 Dec. PMID 32154497